CLINICAL TRIAL: NCT03530514
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, 2-Part Study to Assess the Safety and Tolerability, Pharmacokinetics, And Pharmacodynamics of Single and Multiple Doses of REGN4461 in Healthy Subjects
Brief Title: A Study to Examine the Safety, Tolerability and Biological Effects of REGN4461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: R4461-HV-1794; 2018-000327-14 (EudraCT Number)
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part A: Single dose cohort 1 (Experimental): Cohort 1 will receive a single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 2 (Experimental): Cohort 2 will receive a sequential ascending single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 3 (Experimental): Cohort 3 will receive a sequential ascending single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 4 (Experimental): Cohort 4 will receive a sequential ascending single SC dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 5 (Experimental): Cohort 5 will receive a sequential ascending single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 6 (Experimental): Cohort 6 will receive a sequential ascending single SC dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 7 (Experimental): Cohort 7 will receive a sequential ascending single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 8 (Experimental): Cohort 8 will receive a single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part A: Single dose cohort 9 (Experimental): Cohort 9 will receive a single IV dose of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo
- Part B: Repeated dose cohort 10 (Experimental): Cohort 10 will receive repeated IV or SC doses of REGN4461 or matching placebo
  Interventions: Drug: REGN4461; Drug: Placebo

INTERVENTIONS:
Drug: REGN4461 — REGN4461
Drug: Placebo — Placebo-matching REGN4461

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of REGN4461 in healthy participants. The secondary objectives of the study are to:

* Characterize the Pharmacokinetic (PK) profile of single and repeated doses of REGN4461 and evaluate the effects of baseline covariates on PK profile
* Estimate the effects of repeated doses of REGN4461 on body weight over 12 weeks in overweight and obese participants
* Assess the effects of repeated doses of REGN4461 on ad lib energy intake in overweight and obese participants
* Evaluate the effects of single and repeated doses of REGN4461 on soluble forms of lipid-regulating proteins levels over time
* Assess the immunogenicity of single and repeated doses of REGN4461

DETAILED DESCRIPTION:
This is a 2-part study of the safety, tolerability, PK and pharmacodynamic (PD) of single and repeated doses of REGN4461 in healthy participants. In Part A, healthy lean or overweight participants will be enrolled to evaluate the safety, tolerability, PK, and PD of single ascending intravenous (IV) and subcutaneous (SC) doses. Interim PK and safety information from Part A will be used to select the dose level, frequency, and mode of administration (IV or SC) for repeat dosing in Part B. In Part B, overweight/obese participants with body mass index (BMI) 25-40 kg/m2 will be enrolled to evaluate the safety, tolerability, PK, and PD of repeated doses of REGN4461 in 4 distinct cohorts defined by baseline leptin levels.

ELIGIBILITY:
Key Inclusion Criteria

Part A:

* Males and females 18 to 50 years of age, inclusive
* Body mass index (BMI) from 18.5 to <30.0 kg/m^2
* Participant is judged by the investigator to be in good health and free from major comorbidities based on medical history, physical examination, laboratory safety tests performed at screening and/or prior to administration of initial dose of study drug

Part B:

* Males and females 18 to 65 years of age, inclusive
* Have a body mass index (BMI) from 25.0 to 40.0 kg/m^2
* Participant is judged by the investigator to be free from major comorbidities based upon medical history, physical examination, laboratory safety tests performed at screening and/or prior to administration of initial dose of study drug. Participants can have a history of mild hyperlipidemia and/or mild hypertension but should be on stable doses of lipid lowering or blood pressure lowering medicines for at least 2 months prior to screening

Key Exclusion Criteria

Part A:

* History of type 1 or 2 diabetes or prediabetes or with fasting blood glucose (FBG) at screening ≥ 100mg/dL or with HbA1c at screening of ≥ 5.7%.
* Fasting LDL-C ≥ 130mg/dL, TG ≥ 250 mg/dL

Part B:

* History of type 1 or 2 diabetes or with FBG at screening ≥ 126 mg/dL or with HbA1c at screening of ≥ 6.5%. A diagnosis of "pre-diabetes" is allowed.
* Fasting LDL-C ≥ 160 or TG ≥ 500 mg/dL

Key Exclusion Criteria (Parts A and B):

* Hospitalization (ie, >24 hours) for any reason within 60 days of the screening visit
* History of hypothalamic amenorrhea or lipodystrophy.
* Change in body weight of more than 5% over the past 3 months prior to screening.
* Previous history of bariatric procedures for obesity (eg, sleeve gastrectomy, gastric bypass, banding, etc).
* Procedures for weight reduction (eg, liposuction) or body contouring in the past 6 months.
* Treatment with medications for (over-the-counter [OTC] or prescribed) weight loss (eg, lorcaserin, phentermine/topiramate, naltrexone HCl/bupropion HCl, liraglutide) in the past 3 months.
* History of major psychiatric disorders, eating disorders (eg, bulimia, anorexia).
* Current cigarette smoker or former smoker (cigarettes or e-cigarettes) who stopped smoking within 3 months prior to screening.
* History of recreational drug (including marijuana) or alcohol abuse (>2 drinks per day) within a year prior to the screening visit.
* History of hepatitis B infection or a positive hepatitis B surface antigen (HbsAg+) at screening
* History of HIV infection or HIV seropositive at the screening visit.
* History of hepatitis C infection or positive hepatitis C antibody test result at screening.
* Pregnant or breastfeeding women.

Note: Other inclusion/ exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) | Up to week 27

SECONDARY OUTCOMES:
Concentrations of REGN4461 in serum over time | Up to week 27
Percent change from baseline to week 12 in body weight in overweight or obese participants | Baseline to week 12
Absolute change from baseline to week 12 in body weight in overweight or obese participants | Baseline to week 12
Change from baseline in caloric intake in response to standardized meals in overweight or obese participants | Baseline to week 12
Change in lipid-regulating protein levels over time after single doses of REGN4461 | Up to week 16
Change in lipid-regulating protein levels over time after repeated doses of REGN4461 | Up to week 27
Incidence of anti-drug antibodies to REGN4461 over time after single doses of REGN4461 | Up to week 16
Incidence of anti-drug antibodies to REGN4461 over time after repeated doses of REGN4461 | Up to week 27
Pharmacokinetic (PK) parameter: Area under curve (AUC) computed from time zero to the time of the last positive concentration (AUClast) | Up to week 27
PK parameter: AUC computed across a dosing interval with length τ (AUCo-τ) | Upt to week 27
PK parameter: peak concentration (Cmax) | Up to week 27
PK parameter: time to Cmax (tmax) | Up to week 27
PK parameter: clearance (CL) | Up to week 27
PK parameter: trough concentration (Ctrough) | Up to week 27

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Investigational Site, Antwerp, Belgium